CLINICAL TRIAL: NCT01652521
Title: Effects of Pleural Effusion Drainage on Respiratory System Mechanics in Mechanically Ventilated Patients, as Measured by Esophageal Balloon.
Brief Title: Effects of Pleural Effusion Drainage on Respiratory System Mechanics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Soroksky Arie, M.D., Wolfson Medical Center
Other Study IDs: 0083-12-WOMC
Record Dates: First submitted 2012-07-23; First posted 2012-07-30 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Pleural Effusion
Keywords: lung compliance; pleural effusion; esophageal pressure
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- candidates for pleural fluid drainage: patients who are candidates for pleural fluid drainage.

SUMMARY:
The effects of pleural drainage on lung mechanics are unknown. Insertion of esophageal balloon will allow us to measure and assess pleural pressure, and thus assess any possible effects of pleural fluid drainage may have on lung mechanics.

DETAILED DESCRIPTION:
Esophageal balloon will be inserted prior to pleural fluid drainage.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated patients with significant pleural fluid documented by CT scan or US.who are candidates for pleural fluid drainage.

Exclusion Criteria:

* Patients with any of the following were excluded from the study. Previous lung or chest wall surgery, previous esophageal surgery, known Achalasia or any other esophageal motility or spasm disorder, presence of chest thoracostomy tube, and any significant chest wall abnormality such as kyphoskoliosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients with significant pleural fluid documented by CT scan or US.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
chest wall and lung compliance | 1 year
  The use of esophageal balloon allows us to partition respiratory system into its components, namely, chest wall and lung compliance. These measurements have not been described so far in patients undergoing pleural fluid drainage. Thus, assessment of esophageal pressure which is a surrogate of pleural pressure will allow us an accurate measurement of the effect of pleural fluid drainage on chest wall and lung mechanics.

SECONDARY OUTCOMES:
oxygenation | 1 year
  We suspect that pleural fluid drainage will be associated with improved chest wall and lung mechanics. If this will be the case, then we expect a concomitant improvement in oxygenation.

CONTACTS AND LOCATIONS:
Overall Officials: Arie Soroksky, MD, Principal Investigator — Wolfson MC
Locations (1):
- Wolfson MC, Holon, Israel

REFERENCES:
- [Background] Brown NE, Zamel N, Aberman A. Changes in pulmonary mechanics and gas exchange following thoracocentesis. Chest. 1978 Nov;74(5):540-2. doi: 10.1378/chest.74.5.540. PMID 738092